CLINICAL TRIAL: NCT00000252
Title: Lack of Acute Tolerance Development to Effects of Nitrous Oxide
Brief Title: Lack of Acute Tolerance Development to Effects of Nitrous Oxide - 4
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-08391-4; R01DA008391 (NIH); R01-08391-4
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Opioid-Related Disorders; Substance-Related Disorders
Keywords: nitrous oxide; acute tolerance; subjective effects; psychomotor; analgesia; healthy volunteer
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders; Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- 0% N2O (Sham Comparator): Subjects will inhale 0% N2O
  Interventions: Drug: 0% N2O
- 10% N2O (Active Comparator): Subjects will inhale 10% N2O
  Interventions: Drug: 10% N2O
- 20% N2O (Active Comparator): Subjects will inhale 20% N2O
  Interventions: Drug: 20% N2O
- 30% N2O (Active Comparator): Subjects will inhale 30% N2O
  Interventions: Drug: 30% N2O
- 40% N2O (Active Comparator): Subjects will inhale 40% N2O
  Interventions: Drug: 40% N2O

INTERVENTIONS:
Drug: 0% N2O
  Arms: 0% N2O
Drug: 10% N2O
  Arms: 10% N2O
Drug: 20% N2O
  Arms: 20% N2O
Drug: 30% N2O
  Arms: 30% N2O
Drug: 40% N2O
  Arms: 40% N2O

SUMMARY:
The purpose of this study is to conduct experiments to examine subjective and reinforcing effects of nitrous oxide. Mood altering and psychomotor effects will be tested on non-drug abusers and preference procedures will be used to assess reinforcing effects. To examine the lack of acute tolerance development to the subjective, cognitive, and psychomotor effects of nitrous oxide in healthy volunteers.

ELIGIBILITY:
Please contact site for information.

Ages: 21 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 1994-06; Primary Completion 1996-06 (Actual); Study Completion 1996-06 (Actual)

PRIMARY OUTCOMES:
Psychomotor performance | During inhalation
  Subjects will undergo psychomotor testing during 120 min inhalation session of each intervention
Cognitive performance | During inhalation
  Subjects will under cognitive testing during 120 minute inhalation session of each intervention

CONTACTS AND LOCATIONS:
Overall Officials: James Zacny, Ph.D., Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Anesthesia & Critical Care, Chicago, Illinois, United States

REFERENCES:
- [Background] Yajnik S, Zacny JP, Young CJ, Lichtor JL, Rupani G, Klafta JM, Coalson DW, Apfelbaum JL. Lack of acute tolerance development to the subjective, cognitive, and psychomotor effects of nitrous oxide in healthy volunteers. Pharmacol Biochem Behav. 1996 Jun;54(2):501-8. doi: 10.1016/0091-3057(95)02278-3. PMID 8743615